CLINICAL TRIAL: NCT06239649
Title: The Effect of RF Genicular Nerve Block Applied in the Preoperative Period on Fast-track Total Knee Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Harun Resit Gungor, Prof. Dr, Pamukkale University
Other Study IDs: 2023PAUOrto
Record Dates: First submitted 2023-12-27; First posted 2024-02-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic
Keywords: Fast-Track Total Knee Arthroplasty; Genicular Nerve Block; Radiofrequency Ablation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TKA with radiofrequency ablation genicular nerve block: TKA with radiofrequency ablation genicular nerve block
  Interventions: Procedure: Genicular nerve Radiofrequency Ablation block
- TKA without nerve block: TKA without radiofrequency ablation genicular nerve block

INTERVENTIONS:
Procedure: Genicular nerve Radiofrequency Ablation block — Genicular nerve Radiofrequency Ablation block
  Groups: TKA with radiofrequency ablation genicular nerve block

SUMMARY:
In our study, investigators plan to compare the preoperative RF and genicular nerve ablation approach in patients who underwent TKA(Total Knee Arthroplasty) using the Fast-Track protocol in terms of meeting postoperative pain, function and early discharge criteria.

DETAILED DESCRIPTION:
One of the most important components of surgery using Fast-Track is the application of effective and well-monitored pain treatment. Post-surgical pain negatively affects the patient's early mobilization. Reduction in pain after TKA(Total Knee Arthroplasty) may not only increase short-term functional results but also increase the patient's overall satisfaction.

Genicular Nerve Radiofrequency Ablation (GNRFA) is a non-surgical treatment increasingly used in patients with advanced knee osteoarthritis. Previous studies have shown this to be an effective and safe method to reduce pain and improve functionality in this patient population.

Neurolysis of genicular nerves with radiofrequency (RF) may be useful to relieve pain and improve both function and quality of life in patients with post-TKA pain.

Investigators thought that reducing the pain of patients who underwent TKA with Fast-track in the postoperative period would contribute to early mobilization and therefore rapid functional recovery. As a result of previous studies, investigators know that genicular nerve neurolysis with RF Ablation in the preoperative period provides a reduction in postoperative pain.

Investigators routinely apply TKA applications in clinic with Fast-Track. In investigators hospital's algology outpatient clinic, genicular nerve RF ablation is routinely performed under USG or fluoroscopy guidance. In investigators study, investigators plan to compare the preoperative RF and genicular nerve ablation approach in patients who underwent TKA using the Fast-Track protocol in terms of meeting postoperative pain, function and early discharge criteria

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40 and 85,
* Being able to understand verbal and written information given in Turkish,
* Being able to speak and understand Turkish,
* Being subjected to unilateral TKA surgery due to the diagnosis of Primary Knee osteoarthritis

Exclusion Criteria:

* Patients planned for revision knee prosthesis surgery,
* Patients previously diagnosed with psychiatric disorders,
* Patients who have undergone major surgery on the extremity where TKA will be applied,
* Patients with comorbid diseases such as rheumatoid arthritis or cancer,
* Patients with a score above 3 according to the American Society of Anesthesiologists (ASA) scoring,
* Patients with neurological diseases that cause functional disability,
* Patients with flexion limitation of more than 45 degrees and extension limitation of more than 20 degrees,
* Patients who have to use hypnotic or anxiolytic drugs regularly,
* Patients with alcohol or drug addiction,
* Patients with bleeding disorders
* Patients with uncontrolled diabetes

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Being between the ages of 40 and 85,
  * Being able to understand verbal and written information given in Turkish,
  * Being able to speak and understand Turkish,
  * Being subjected to unilateral TKA surgery due to the diagnosis of Primary Knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain preoperative | Baseline (preoperatively)
  Visual Analog Scale used to assess pain
Pain postoperative 1 | at postoperative sixth weeks
  Visual Analog Scale used to assess pain
Pain postoperative 2 | at postoperative twelfth weeks
  Visual Analog Scale used to assess pain
Knee Range of Motion preoperative | Baseline (preoperatively)
  Digital goniometer used to assess knee range of motion
Knee Range of Motion postoperative 1 | at postoperative sixth week
  Digital goniometer used to assess knee range of motion
Knee Range of Motion postoperative 2 | at postoperative twelfth week
  Digital goniometer used to assess knee range of motion
Quadriceps muscle strength preoperative | Baseline (preoperatively)
  Quadriceps muscle strength is measured (unit=newton(N)) with hand-held dynamometer
Quadriceps muscle strength postoperative 1 | at postoperative sixth weeks
  Quadriceps muscle strength is measured (unit=newton(N)) with hand-held dynamometer
Quadriceps muscle strength postoperative 2 | at postoperative twelfth week
  Quadriceps muscle strength is measured (unit=newton(N)) with hand-held dynamometer
Patient-reported activity limitations preoperative | Baseline (preoperatively)
  The Western Ontario and McMaster Universities Arthritis Index and Knee injury and Osteoarthritis Outcome Score are used
Patient-reported activity limitations preoperative 1 | at postoperative sixth weeks
  The Western Ontario and McMaster Universities Arthritis Index and Knee injury and Osteoarthritis Outcome Score are used
Patient-reported activity limitations preoperative 2 | at postoperative twelfth week
  The Western Ontario and McMaster Universities Arthritis Index and Knee injury and Osteoarthritis Outcome Score are used
Performance-based activity limitations-preoperative | Baseline (preoperatively)
  30-sec chair-stand test and stair-climb test are used
Performance-based activity limitations-preoperative 1 | at postoperative sixth weeks
  30-sec chair-stand test and stair-climb test are used
Performance-based activity limitations-preoperative 2 | at postoperative twelfth week
  30-sec chair-stand test and stair-climb test are used
Quality of life-preoperative | Baseline (preoperatively)
  Short Form-36 (SF-36) is used
Quality of life-preoperative 1 | at postoperative sixth weeks
  Short Form-36 (SF-36) is used
Quality of life-preoperative 2 | at postoperative twelfth week
  Short Form-36 (SF-36) is used
Length of hospital stay | through study completion, an average of 1 year
  Length of hospital stay is measured beginning from the hospitalization of the patient and ending at discharge of the patients (unit-hours)

SECONDARY OUTCOMES:
Length of operation time | the surgery
  Length of operation time is measured in minutes during the surgery
Amount of blood loss | through study completion, an average of 1 year
  Amount of blood loss is measured from the suction drainage (unit-milliliters)
postoperative component alignments | through study completion, an average of 1 year
  Long leg radiographs of the patients are evaluated postoperatively by using a digital orthopedic templating software-Materialise OrthoView (OrthoView version 7, Materialise HQ, Technologielaan 15 3001 Leuven, Belgium).

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stake S, Agarwal AR, Coombs S, Cohen JS, Golladay GJ, Campbell JC, Thakkar SC. Total Knee Arthroplasty After Genicular Nerve Radiofrequency Ablation: Reduction in Prolonged Opioid Use Without Increased Postsurgical Complications. J Am Acad Orthop Surg Glob Res Rev. 2022 Aug 12;6(8):e22.00125. doi: 10.5435/JAAOSGlobal-D-22-00125. eCollection 2022 Aug 1. PMID 35960987
- [Background] Lloyd JM, Wainwright T, Middleton RG. What is the role of minimally invasive surgery in a fast track hip and knee replacement pathway? Ann R Coll Surg Engl. 2012 Apr;94(3):148-51. doi: 10.1308/003588412X13171221590214. PMID 22507716
- [Background] Sullivan M, Tanzer M, Reardon G, Amirault D, Dunbar M, Stanish W. The role of presurgical expectancies in predicting pain and function one year following total knee arthroplasty. Pain. 2011 Oct;152(10):2287-2293. doi: 10.1016/j.pain.2011.06.014. Epub 2011 Jul 18. PMID 21764515